CLINICAL TRIAL: NCT03187431
Title: Mesenchymal Stem Cell as Therapeutic Modality in Interstitial Pulmonary Fibrosis
Brief Title: Role of Stem Cell Therapy in Interstitial Pulmonary Fibrosis
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Prof. Dr. Aliae AR Mohamed-Hussein, Professor of Pulmonology, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AssiutU4
Record Dates: First submitted 2017-04-11; First posted 2017-06-15 (Actual); Last update posted 2017-06-15 (Actual); Status verified 2017-06

CONDITIONS: Stem Cell Transplant Complications
Keywords: Stem cell; Therapy; IPF

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IPF patients (Experimental): autologous bone marrow mesenchymal stem cells
  Interventions: Biological: autologous bone marrow mesenchymal stem cells

INTERVENTIONS:
Biological: autologous bone marrow mesenchymal stem cells — intravenous infusion

SUMMARY:
Currently, the application status of MSCs as treatment modalities in IPF is still in its infancy and remains exploratory. Although a number of safety and efficacy clinical trials of MSCs as therapeutic options in immune-mediated and cardiac diseases have already been published with tantalizing results, to our disappointment, pulmonary and critical care medicine have traditionally lagged behind other therapeutic and research fields including hematology, gastroenterology and cardiology in translational studies of the use of reparative cells

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 75 years (both inclusive)
* high-resolution computed tomography (HRCT) scan that is very suggestive or consistent with a probable diagnosis of usual interstitial pneumonia.
* Bronchoalveolar lavage must be performed at any time before inclusion and must have failed to show features supporting alternative diagnoses.
* The duration of the disease should be more than three months, and bibasilar inspiratory crackles should be present.
* dyspnea score of at least 2 on a scale of 0 (minimum) to 10 (maximum).
* FVC > 50% of the predicted normal value and DLco > 35% of the predicted value.
* Patients under treatment with n-acetylcysteine or pirfenidone should discontinue drug and enter a wash-out period for at least 6 weeks prior study enrolment.

Exclusion Criteria:

* FVC < 50% predicted normal value and DLCO < 35%predicted normal value.
* lung cancer or with an evidence of active malignancyfor at least 5 years.
* uncontrolled heart failure.
* renal failure
* hepatic failure,
* neurological abnormalities including stroke and myasthenia Gravis
* Anti-coagulants therapy.
* Active infections.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2017-12-11 (Estimated); Primary Completion 2018-10-01 (Estimated); Study Completion 2018-12-01 (Estimated)

PRIMARY OUTCOMES:
number of participants with treatment related side effects as infection, allergic reaction, disease acute exacerbation, and ectopic tissue formation | 6 months
  safety and side effects

SECONDARY OUTCOMES:
Post therapy diffusing capacity of CO% (DLCO)predicted | 6-12 months
  Efficacy of procedure
post therapy forced vital capacity (FVC)% predicted. | 6-12 months
  efficacy of the procedure

IPD SHARING:
Plan to Share IPD: No